CLINICAL TRIAL: NCT03361072
Title: The Effect of Per Oral Immunotherapy Treatment in Severe IgE Mediated Milk, Peanut and Egg Allergy in Adults
Brief Title: The Effect of Per Oral Immunotherapy in Severe Milk, Peanut and Egg Allergy in Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Paula Kauppi, MD, PhD, MD, PhD, Chief Specialist, Helsinki University Central Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUS/486/2017
Record Dates: First submitted 2017-08-11; First posted 2017-12-04 (Actual); Results first posted 2025-05-09 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Food Allergy
Keywords: oral immunotherapy; milk; peanut; egg; adult
MeSH Terms: conditions — Food Hypersensitivity | interventions — Immunotherapy

STUDY DESIGN:
Intervention Model Description: Prospective open label study on oral immunotherapy with either milk, or peanut or egg white food products.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Milk allergy (Experimental): Milk oral immunotherapy intervention for milk allergy
  Interventions: Dietary Supplement: Oral immunotherapy
- Peanut allergy (Experimental): Peanut oral immunotherapy intervention for peanut allergy
  Interventions: Dietary Supplement: Oral immunotherapy
- Egg allergy (Experimental): Egg oral immunotherapy intervention for egg allergy
  Interventions: Dietary Supplement: Oral immunotherapy

INTERVENTIONS:
Dietary Supplement: Oral immunotherapy — Milk, peanut or egg oral immunotherapy

SUMMARY:
The aim is to analyse the results of per oral immunotherapy treatment in severe milk, peanut or egg allergy in adults. This is the second part of the oral immunotherapy study in adults at Skin and Allergy Hospital. The diagnosis of food allergy is verified with positive history, skin prick tests, egg and milk allergen specific IgE (immunoglobulin E) antibodies. In addition, food allergy is verified with an open label (milk allergy) or blind (peanut and egg allergy) allergen specific challenge test. OIT (oral immunotherapy) is performed according to a detailed plan. Lung function parameters are followed before OIT and and a year after OIT.

DETAILED DESCRIPTION:
30 patients with milk allergy (at least 18 year olds), 30 patients with peanut allergy and 30 patients with egg allergy are treated with OIT. The diagnosis of food allergy is verified with positive history, skin prick test, egg and milk allergen specific IgE antibodies. In addition, food allergy is verified with an open label (milk allergy) or blind (peanut and egg allergy) allergen specific challenge test. Quality of life, anxiety and patient history data is collected by questionnaires. All the patients undergo a spirometry with a bronchodilatator test, exhaled nitric oxide test and a methacholine challenge before and a year after oral immunotherapy. All the patients undergoing oral immunotherapy are prescribed with emergency medication such as antihistamine tablets, prednisolon tablets (40mg for three days in adults), epinephrine autoinjector (300 µg per dose) and salbutamol or terbutaline inhalator.

ELIGIBILITY:
Inclusion Criteria:

* severe milk, peanut or egg allergy verified with positive symptom history, skin prick tests and serum IgE tests and a challenge test

Exclusion Criteria:

* instable cerebrovascular or heart disease, active autoimmune disease or cancer, or current use of betablockers.
* poorly controlled asthma or FEV1 < 70% (FEV1< -2SD)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-08-03 (Actual); Primary Completion 2023-03-11 (Actual); Study Completion 2023-03-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paula Kauppi, MD, PhD, Principal Investigator — Helsinki University Central Hospital
Locations (1):
- Helsinki University Central Hospital, Helsinki, Finland

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Milk Allergy | Peanut Allergy | Egg Allergy
Started | 12 | 14 | 4
Completed | 8 | 5 | 2
Not Completed | 4 | 9 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Milk Allergy | Peanut Allergy | Egg Allergy | Total
Number analyzed (Participants) | 12 | 14 | 4 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 12 | 14 | 4 | 30
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.8 (12.5) | 29.6 (11.0) | 25.3 (20.5) | 31.1 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 9 | 4 | 24
  Male | 1 | 5 | 0 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 12 | 14 | 4 | 30
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Finland | 12 | 14 | 4 | 30

OUTCOME MEASURES:

1. Primary Outcome: Desensitisation
Description: Increase in tolerated dose (that is no symptoms if accidental exposure) of food compared to the pre-OIT, number of participants
Time Frame: 1 year, through study completion
Measure: Count of Participants; unit: Participants
Arm/Group | Milk Allergy | Peanut Allergy | Egg Allergy
Number analyzed (Participants) | 12 | 14 | 4
Participants | 7 | 5 | 2

2. Secondary Outcome: Worries Associated With Food Allergy
Description: Quality of life and reported concerns and worries associated with food allergy using a VAS scale (visual analogue scale) from 0 (no worries) to 100 mm (maximal worries) before OIT and at one year after OIT
Time Frame: 1 year, through study completion
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Milk Allergy | Peanut Allergy | Egg Allergy
Number analyzed (Participants) | 10 | 7 | 4
score on a scale
  Before OIT (VAS) | 77.7 (19.2) | 69.7 (12.4) | 61.0 (13.0)
  After OIT, at one year (VAS) | 79.00 (5.6) | 39.5 (19.1) | 25.0 (0.0)

3. Other Pre Specified Outcome: Number of Participants With Treatment-related Adverse Events
Description: Follow-up of safety of OIT, Number of participants with treatment-related adverse events
Time Frame: 1 year, through study completion
Measure: Count of Participants; unit: Participants
Arm/Group | Milk Allergy | Peanut Allergy | Egg Allergy
Number analyzed (Participants) | 12 | 14 | 4
Participants | 12 | 14 | 4

4. Other Pre Specified Outcome: Decrease in Allergen Specific IgE Values
Description: Allergen specific IgE values before OIT and after OIT (kU/l)
Time Frame: 1 year, through study completion
Population: S-IgE milk for milk allergy, S-IgE peanut for peanut allergy, S-IgE egg white for egg allergy
Measure: Mean (Standard Deviation); unit: kU/l
Arm/Group | Milk Allergy | Peanut Allergy | Egg Allergy
Number analyzed (Participants) | 11 | 14 | 4
kU/l
  IgE pre OIT | 100.7 (112.4) | 88.4 (212.8) | 81.3 (81.1)
  IgE post OIT | 4.1 (5.4) | 26.4 (27.2) | 27.6 (3.3)

ADVERSE EVENTS:
Time Frame: OIT after two years post start
Description: OIT after two years post start
Arm/Group | Milk Allergy | Peanut Allergy | Egg Allergy
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/14 | 0/4
Serious Adverse Events (participants affected / at risk) | 4/12 | 2/14 | 0/4
Other Adverse Events (participants affected / at risk) | 8/12 | 12/14 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Milk Allergy (N=12) | Peanut Allergy (N=14) | Egg Allergy (N=4)
Allergic reaction (Skin and subcutaneous tissue disorders) | 4 (4) | 2 (2) | 0 (0) — EpiPen usage or emergency visit because of OIT and allergy reaction
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Milk Allergy (N=12) | Peanut Allergy (N=14) | Egg Allergy (N=4)
Local itching (Skin and subcutaneous tissue disorders) | 8 (8) | 12 (12) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigators will postpone single-site publications until after publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-07): https://cdn.clinicaltrials.gov/large-docs/72/NCT03361072/Prot_SAP_000.pdf